CLINICAL TRIAL: NCT03970070
Title: Perioperative Ostomy Self-Management Telehealth (Periop-OSMT) for Cancer Patients and Family Caregivers
Brief Title: Perioperative Ostomy Self-Management Telehealth for Cancer Patients and Family Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18327; NCI-2019-02385 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18327 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2019-05-01; First posted 2019-05-31 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health service research (Periop-OSMT) (Experimental): Patients and/or support persons/family caregivers complete Periop-OSMT session in-person or via telephone over 20-40 minutes before surgery and before hospital discharge and group telehealth session over 1.5-2 hours at weeks 1-3, 4, 5, 6, and 7 post discharge
  Interventions: Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Informational Intervention — Complete Perioperative Ostomy Self-Management Telehealth program
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well Perioperative Ostomy Self-Management Telehealth (Periop-OSMT) provides patients and their caregivers information about ostomy and ostomy care. Periop-OSMT may help to understand patient preparedness to do ostomy self-care, confidence in doing ostomy self-care, knowledge of ostomy self-care, quality of life, mood, use of medical services, and financial burden.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the feasibility and acceptability of the Periop-OSMT as measured by the percentage of patients and support persons/family caregivers (FCGs) who agree to participate; complete >= 80% of the intervention; and report satisfaction with the intervention (through structured exit interviews).

SECONDARY OBJECTIVES:

I. Examine the patterns and trajectories for patient outcomes pre- and post-intervention, including patient activation, self-efficacy, ostomy-related knowledge, health related quality of life (HRQOL), medical care utilization, and financial burden.

II. Examine patterns and trajectories for support person/FCG outcomes pre- and post-intervention, including quality of life (QOL).

III. Using qualitative methods, evaluate the acceptability of the intervention as reported by participants.

OUTLINE:

Patients and/or support persons/family caregivers complete Periop-OSMT session in-person or via telephone over 20-40 minutes before surgery and before hospital discharge, and group telehealth session over 1.5-2 hours at weeks 1-3, 4, 5, 6, and 7 post discharge.

After completion of study intervention, participants are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Scheduled to undergo a surgical procedure that includes the creation of an intestinal stoma (fecal or urinary).
* PATIENT: Able to read and understand English.
* PATIENT: Patients scheduled for temporary ostomy procedures
* SUPPORT PERSON/FCG: Family member/friend identified by the patient as the primary caregiver before and after surgery.
* SUPPORT PERSON/FCG: Able to read and understand English.
* Patients with all stages of disease are eligible for the study.
* The study is open to anyone regardless of gender or ethnicity. Efforts are made to extend the accrual to a representative population.

Exclusion Criteria:

* Subjects, who in the opinion of the principal investigator (PI), may not be able to comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Patient and family caregiver (FCG) participation | Up to 24 months
  Assessed by ratio of eligible participants (patient and FCGs) to those enrolled and those who decline participation, reasons for non-participation, number of scheduled study encounters completed, attrition rate between pre- and post-intervention, reasons for attrition/dropout, level of intervention participation including the total number of sessions, number of sessions completed without break-offs, number of break-offs, length (minutes) of sessions, and the ratio of all participants to those who completed >= 80% of the study.

SECONDARY OUTCOMES:
Patient reported outcomes | Up to 6 months post-discharge
  Will be examined pre- and post-intervention, including patient activation, self-efficacy, ostomy-related knowledge, health related quality of life, medical care utilization, and financial burden. Descriptive statistics will be summarized using validated scoring procedures. The data will be used to assess descriptively the trajectory and patterns of outcomes before and after the intervention.
Support person/FCG reported outcomes | Up to 6 months post-discharge
  Will be examined pre- and post-intervention, including quality of life. Descriptive statistics will be summarized using validated scoring procedures. The data will be used to assess descriptively the trajectory and patterns of outcomes before and after the intervention.
Acceptability of Perioperative Ostomy Self-Management Telehealth | Up to 24 months
  Acceptability will be assessed through qualitative data analysis using the conventional content analysis approach. Data from the tape-recorded interviews are transcribed and analyzed using HyperRESEARCH software. Transcripts will be imported for the development of analytic categories, data coding, and review of coded data. All data will be read repeatedly to achieve immersion and obtain a sense of the whole. Then, data will be read word by word to derive codes. Codes will be then sorted into themes based on links and relationship. Separate investigators will conduct a final validation review of the codes and themes to ensure consistency and clarity across all qualitative data. Data discordantly coded will be discussed for refinement and consensus purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - City of Hope Medical Center, Duarte, California
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania